CLINICAL TRIAL: NCT04940403
Title: BurtVision™ for Arm Rehabilitation in Chronic Stroke Survivors: a Comparison of Unimanual vs. Unimanual and Bimanual Tasks During Robot-assisted Arm Training
Brief Title: BurtVision™ for Arm Rehabilitation in Chronic Stroke Survivors:
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Associate Professor, HMS and Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P001807
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to either 1) manual robot-assisted upper-limb rehabilitation, and 2) unimanual+bimanual robot-assisted upper-limb rehabilitation
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Unimanual robot-assisted upper-limb rehabilitation (Active Comparator): Participants randomized to this arm of the study will undergo 18 one-hour sessions of robot-assisted upper-limb rehabilitation. During the sessions, study participants will only train their hemiparetic arm (unimanual tasks only).
  Interventions: Device: Burt
- Bimanual robot-assisted upper-limb rehabilitation (Experimental): Participants randomized to this arm of the study will undergo 18 one-hour sessions of robot-assisted upper-limb rehabilitation. During the sessions, study participants will train their hemiparetic arm as well as interacting with the contralateral arm for bimanual tasks (unimanual + bimanual tasks).
  Interventions: Device: Burt + BurtVision

INTERVENTIONS:
Device: Burt — 18 one-hour sessions of unimanual upper-limb tasks during robot-assisted training with the Burt.
  Arms: Unimanual robot-assisted upper-limb rehabilitation
Device: Burt + BurtVision — 18 one-hour sessions of combination of unimanual and bimanual upper-limb tasks during robot-assisted training with the BurtVision.
  Arms: Bimanual robot-assisted upper-limb rehabilitation

SUMMARY:
The focus of this study is to perform a preliminary assessment of the efficacy of the BurtVision system. While the Burt robotic-arm assists the patient's upper-limb in their movements, BurtVision will allow the patient to perform unimanual and bimanual activities while leveraging augmented reality games. The investigators will compare clinical outcomes when the BurtVisions ystem is used for training solely relying on unimanual tasks vs. when it is used for training relying on both unimanual and bimanual tasks.

DETAILED DESCRIPTION:
The proposed study is a single-blinded randomized clinical trial to evaluate the effect of using the BurtVistion on motor gains after robot-assisted upper-limb. Study participants (stroke survivors) will be recruited at the Spaulding Rehabilitation Hospital - Boston. Subjects will be randomly assigned to one of the two different groups: unimanual or unimanual + bimanual arm therapy using a block-randomized allocation procedure to ensure important covariates, such as baseline Fugl-Meyer Assessment of the Upper Extremity (FMA-UE) scores and chronicity, are balanced between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-80 years old;
2. Unilateral ischemic or hemorrhagic stroke at least 6 months and no more than 5 years prior to study enrollment;
3. Upper extremity hemiparesis as characterized by initial scores on upper limb subtest of the Fugl-Meyer Assessment (FMA-UE) between 12 and 40;
4. Some active pro-supination range of motion;
5. Some active metacarpal-phalangeal joint in the hemiparetic hand;
6. Intact cognitive function to understand the robotic therapy procedures (MMSE>23 and able to follow 3 step command) during initial evaluation visit;

Exclusion Criteria:

1. Undergoing upper-limb rehabilitation therapy during the period of the study.
2. Severe spasticity (defined as a Modified Ashworth scale score of 3 or more) that would prevent safe use of the robotic system;
3. Visual impairments as assessed by the NIH Stroke Scale Visual Field subscale (only subjects with no visual loss will participate in the study); or hemispatial neglect that would impair the subject's ability to play the interactive games (as assessed with the line bisection test);
4. Severe proprioceptive deficits that impair the ability to process haptic or visual feedback, as assessed by physical examination during screening;
5. Communication impairments such aphasia that impair the subject's ability of providing feedback (as reported by a physician in his/her medical record);
6. Individuals with open wounds or recent fracture (<3 months) in the upper extremity, fragile skin or active infection;
7. Upper-extremity orthopedic injuries or severe pain resulting in movement limitations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Motor Activity Log- Amount of Use | Data will be collected at baseline and at 7-8 weeks
  Self-reported measures of upper extremity activity performance in daily life (amount of use)

SECONDARY OUTCOMES:
Fugl-Meyer Assessment, Upper-Extremity portion | Data will be collected at baseline and at 7-8 weeks
  Assessment of the severity of upper-limb motor impairments
Wolf Motor Function Test | Data will be collected at baseline and at 7-8 weeks
  Assessment of arm functional limitations
Stroke Impact Scale | Data will be collected at baseline and at 7-8 weeks
  Self-reported measure of quality of life after stroke
Motor Activity Log- Quality of Use | Data will be collected at baseline and at 7-8 weeks
  Self-reported measures of upper extremity activity performance in daily life (quality of use)
Upper-Extremity Accelerometry | Data will be collected at baseline and at 7-8 weeks
  Amount of arm use over 72 hours recording with wrist-worn sensors

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Harvard Medical School, Spaulding Rehabilitation Hospital

IPD SHARING:
Plan to Share IPD: No